CLINICAL TRIAL: NCT06758622
Title: Multicenter Analysis of Morbidity, Mortality and Medical Care in Neonates At the Isidro Ayora Gynecological-Obstetric Hospital, the Calderón General Teaching Hospital and the Nueva Aurora Luz Elena Arismendi Pediatric Gynecological-Obstetric Hospital, January 2008-June 2024
Brief Title: Analysis on the Health of Newborns in Three Hospitals, 2008-2024
Status: Active, not recruiting | Type: Observational
Sponsor: HOSPITAL GINECO OBSTETRICO ISIDRO AYORA (Other)
Collaborators: Universidad Central del Ecuador (Other)
Responsible Party: Principal Investigator, Santiago Vasco-Morales, MEDICO PEDIATRA, HOSPITAL GINECO OBSTETRICO ISIDRO AYORA
Other Study IDs: CEISH-HGDC-2024-007
Record Dates: First submitted 2024-12-20; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Neonatal Morbidity and Mortality; Intrauterine Growth Disorders (IUGR and Macrosomia); Prematurity Complications; Neonatal Infections
Keywords: Neonatal Mortality; Neonatal Morbidity; Infant, Low Birth Weight
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Definition: This group includes neonates admitted to HGOIA, HGDC, and HGONA between January 2008 and

SUMMARY:
The objective of this observational study is to analyze the factors associated with neonatal morbidity and mortality in three hospitals in Quito, Ecuador, from January 2022 to December 2023. The primary question to be addressed is:

What perinatal factors are associated with neonatal morbidity and mortality in neonates admitted to HGOIA, HGDC, and HGONA hospitals?

The participants will be neonates whose complete medical records are registered in the Perinatal Information System (SIP) and the Maternal-Perinatal Clinical Record (HCMP) databases during the study period. Data will be retrospectively collected from the mentioned databases, evaluating variables such as birth weight, gestational age, congenital anomalies, neonatal complications, and maternal factors such as age and medical conditions.

The analysis will include prevalence calculations, variable associations through logistic regression, and the development of neonatal growth curves. Statistical software such as R will be used for data analysis, and the results will be compared to national and international standards.

DETAILED DESCRIPTION:
Detailed Description of the Study

This retrospective observational study aims to analyze the factors associated with neonatal morbidity and mortality in three hospitals in Quito, Ecuador: the Hospital Gineco Obstétrico Isidro Ayora (HGOIA), the Hospital General Docente de Calderón (HGDC), and the Hospital Gineco Obstétrico Pediátrico de Nueva Aurora Luz Elena Arismendi (HGONA). The study spans the period from January 2022 to December 2023 and utilizes secondary data obtained from the Perinatal Information System (SIP) and the Maternal-Perinatal Clinical Record (HCMP).

Background and Rationale:

The analysis of perinatal factors related to neonatal morbidity and mortality is crucial to improving neonatal care standards and reducing mortality rates. According to the Ecuadorian Ministry of Public Health, the main causes of neonatal mortality in 2020 included prematurity, respiratory distress syndrome, and congenital anomalies, among others. This study seeks to identify and quantify risk and protective factors in the neonatal population admitted to the three mentioned hospitals, enabling the design of more effective interventions.

Methodology:

A cross-sectional design with retrospective data collection will be utilized. The study participants will include all neonates recorded in the SIP and HCMP databases during the specified period. Data will encompass perinatal variables such as birth weight, gestational age, congenital anomalies, neonatal complications, and maternal conditions (e.g., age, comorbidities).

Procedures:

Data Collection:

Extraction of relevant information from the SIP and HCMP databases. Identification and removal of duplicate or incomplete records. Organization of variables using an operationalization chart detailing dimensions, indicators, and measurement scales.

Statistical Analysis:

Bivariate and multivariate analyses will be conducted using logistic regression models to evaluate associations between variables.

Odds ratios (OR) with 95% confidence intervals will be calculated. Neonatal growth curves stratified by sex and gestational age will be generated. R software will be used for all statistical analyses.

Expected Outcomes:

Identification of risk and protective factors associated with neonatal morbidity and mortality.

Characterization of intrauterine growth disorders, prematurity complications, and congenital anomalies in the studied population.

Comparison of indicators across the three hospitals to identify significant differences and design improvement strategies.

Limitations:

Potential biases are anticipated, including errors in clinical record documentation and incomplete data. These limitations will be addressed through thorough data cleaning and exclusion of inconsistent records.

Expected Impact:

The findings will contribute to the development of evidence-based neonatal clinical care protocols and guidelines, aiming to reduce morbidity and mortality rates in participating hospitals and serve as a model for other institutions in the country.

ELIGIBILITY:
Inclusion Criteria:

Neonates registered in the Perinatal Information System or the Maternal-Perinatal Clinical Record during the study period (January 2022 to December 2023).

Neonates born in the participating hospitals: Hospital Gineco Obstétrico Isidro Ayora, Hospital General Docente de Calderón, and Hospital Gineco Obstétrico Pediátrico de Nueva Aurora Luz Elena Arismendi.

Perinatal medical records with complete data, including information on birth weight, gestational age, neonatal complications, and maternal conditions.

Exclusion Criteria:

Neonates with incomplete or inconsistent clinical records in the Perinatal Information System or the Maternal-Perinatal Clinical Record.

Perinatal medical records missing key information, such as discharge diagnoses, gestational age, or birth weight.

Neonates born outside the participating institutions during the study period.

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population consists of neonates born between January 2022 and December 2023 at three hospitals in Quito, Ecuador: Hospital Gineco Obstétrico Isidro Ayora, Hospital General Docente de Calderón, and Hospital Gineco Obstétrico Pediátrico de Nueva Aurora Luz Elena Arismendi. These neonates must have complete perinatal medical records documented in the Perinatal Information System or the Maternal-Perinatal Clinical Record.
  The population includes neonates with varying birth weights, gestational ages, and neonatal complications, as well as their associated maternal conditions, such as age, comorbidities, and pregnancy outcomes. The study focuses on analyzing the prevalence of morbidity and mortality, growth disorders (low birth weight and macrosomia), prematurity-related complications, and adherence to neonatal care interventions like the Kangaroo Mother Care program and Human Milk Bank services.
Sampling Method: Non-Probability Sample
Enrollment: 40000 (Actual)
Dates: Start 2024-11-12 (Actual); Primary Completion 2025-11-12 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Neonatal Morbidity and Mortality Rate | 14 years
  Definition: Proportion of neonates experiencing morbidity (severe diseases or complications) or mortality within the first 28 days of life.
  Method of Measurement: Calculation of rates and proportions using Perinatal Information System and Maternal perinatal medical records.
  Unit of Measure: Percentage (%) per 1000 live births. Time Frame: From birth to 28 days of life.

SECONDARY OUTCOMES:
Prevalence of Intrauterine Growth Disorders (Low Birth Weight and Macrosomia) | 14 years
  Definition: Proportion of neonates born with birth weight below 2500 grams (low birth weight) or over 4000 grams (macrosomia).
  Method of Measurement: Analysis of birth weight data using Perinatal Information System and Maternal perinatal medical records.
  Unit of Measure: Percentage (%). Time Frame: At birth.
Incidence of Prematurity-Related Complications | 14 years
  Definition: Frequency of complications such as bronchopulmonary dysplasia, retinopathy of prematurity, and intraventricular hemorrhage.
  Method of Measurement: Identification of diagnoses in clinical records. Unit of Measure: Percentage (%). Time Frame: From birth to 28 days of life.
Comparison of Indicators Across Hospitals | 14 years
  Definition: Significant differences in morbidity, mortality, and complication rates among the three hospitals.
  Method of Measurement: Multivariate statistical analysis. Unit of Measure: Odds ratio (OR) with 95% confidence intervals. Time Frame: Entire study period.

CONTACTS AND LOCATIONS:
Overall Officials: Elina Yanez Valencia, Neonatologa, Study Director — Hospital Docente de Calderon; Monica Diaz Torres, Neonatologa, Principal Investigator — Hospital Gineco Obstétrico Pediátrico de Nueva Aurora Luz Elena Arismendi
Locations (1):
- Hospital Gineco Obstétrico Isidro Ayora, Quito, Pichincha, Ecuador

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosero-Quintana MD, Vasco-Morales S, Benalcazar-Sanmartin K, Salazar-Congacha LP, Toapanta-Pinta PC. Frequency of episiotomy practice in an institution in Quito, Ecuador 2009-2022. Rev Colomb Obstet Ginecol. 2024 Jul 9;75(2):4216. doi: 10.18597/rcog.4216. English, Spanish. PMID 39470265
- See also: Related Info — https://www.medrxiv.org/content/10.1101/2024.06.09.24307243v1